CLINICAL TRIAL: NCT07193901
Title: A Randomized, Double-blind, Placebo-controlled Phase Il Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Characteristics of (R)-Ketamine Hydrochloride Nasal Spray in Patients With Depression and Acute Suicidal Ideation or Behavior
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Characteristics of (R)-Ketamine Hydrochloride Nasal Spray in Patients With Depression and Acute Suicidal Ideation or Behavior
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Purity Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRT042-II-01
Record Dates: First submitted 2025-09-01; First posted 2025-09-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder (MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose PRT042 nasal spray (Experimental)
  Interventions: Drug: Low Dose PRT042 nasal spray
- median Dose PRT042 nasal spray (Experimental)
  Interventions: Drug: median Dose PRT042 nasal spray
- high Dose PRT042 nasal spray (Experimental)
  Interventions: Drug: high dose PRT042 nasal spray
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Low Dose PRT042 nasal spray — two times a week, for 4 weeks
  Arms: Low Dose PRT042 nasal spray
Drug: median Dose PRT042 nasal spray — two times a week, for 4 weeks
  Arms: median Dose PRT042 nasal spray
Drug: high dose PRT042 nasal spray — two times a week, for 4 weeks
  Arms: high Dose PRT042 nasal spray
Drug: placebo — two times a week, for 4 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to learn about:

* To evaluate the efficacy of PRT-042 nasal spray for the Rapid Reduction of the depressive symptoms in adults with major depressive disorder (MDD) with acute suicidal ideation or behavior
* To evaluate the safety and pharmacokinetic (PK) characteristics after multiple dose of PRT-042 nasal spray in adults with major depressive disorder (MDD) with acute suicidal ideation or behavior

ELIGIBILITY:
Inclusion Criteria:

1. Participant must meet Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) diagnostic criteria for Major Depressive Disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Mini International Psychiatric Interview (MINI) .
2. Participants must have current suicidal ideation with intent, confirmed by a "Yes" response to Question B3 [Think (even momentarily) about harming or of hurting or of injuring yourself: with at least some intent or awareness that you might die as a result; or think about suicide (ie, about killing yourself)?] and Question B10 [Intend to act on thoughts of killing yourself?] obtained from the MINI.
3. Participant has a Montgomery Asberg Depression Rating Scale (MADRS) total score of greater than (≥) 28 and the score for item 10"suicide ideation" of greater than (≥) 3 predose on Day 1

Exclusion Criteria:

1. Participant has a current DSM-5 diagnosis of bipolar (or related disorders), antisocial personality disorder, or obsessive compulsive disorder.
2. Participant has a current clinical diagnosis of autism, dementia, or intellectual disability.
3. Participant has a current or prior DSM-5 diagnosis of a psychotic disorder, or MDD with psychotic features .
4. Participant meets the DSM-5 severity criteria for moderate or severe substance or alcohol use disorder, within the 6 months before screening
5. Participant has a current or prior diagnosis of a reatment resistant depression
6. Any nasal conditions or diseases that, in the investigator's judgment, may significantly affect the administration or absorption of a nasal product.
7. Participant has a history of malignancy within 5 years before screening
8. Pregnant or breastfeeding women, or those with a positive pregnancy test result during screening.
9. Previous participation in another clinical trial and receiving the investigational drug within 3 months prior to dosing.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at 24 Hours After the First Dose (Day 2) | Baseline (Day 1, predose) and 24 hours first post dose (Day 2)
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Change From Baseline in Montgomery Asberg Depression Rating Scale Total Score During Double-blind Phase | Days 1 (4 hours postdose), 4, 8, 11, 15, 18, 22 and Day 25
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Number of Participants who Achieved Response （≥50% decrease from baseline MADRS total score）Through the Double-blind Phase | Days 1 (4 hours postdose),2, 4, 8, 11, 15, 18, 22 and Day 25
Number of Participants Who Achieved Remission (MADRS Total Score Less Than or Equal to [<=] 12) Through the Double-blind Phase | Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and Day 25
5. Change From Baseline in Clinical Global Impression- Severity of Suicidality-Revised (CGI-SS-R) During Double-blind Phase | Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and Day 25
  CGI-SS-R was derived from the Clinical Global Impression Severity Scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participants illness. The CGI-SS-R rating is scored on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants). A higher score indicates a more severe condition and a reduction in score indicates improvement (that is, lower severity of suicidality).
Number of Participants Who Achieved Resolution of Suicidality (CGI-SS-R Score of 0 or 1) Through Double-blind Phase | up to Day 25
Change From Baseline in Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) Scale Total Score During Double-blind Phase | Days 1 (4 hours postdose), 2, 4, 8, 11, 15, 18, 22 and Day 25
  The CGI-SR-I is a scale summarizing the clinician's best assessment of the likelihood that the participant will attempt suicide in the next 7 days. The CGI-SR-I rating is scored on a 7-point scale: where' 0 (no imminent suicide risk); 1 (minimal imminent suicide risk), 2 (mild imminent suicide risk), 3 (moderate imminent suicide risk), 4 (marked imminent suicide risk), 5 (severely imminent suicide risk), 6 (extreme imminent suicide risk). Higher score indicates a more severe condition. Negative change in score indicates improvement.
8. Change From Baseline in Beck Hopelessness Scale (BHS) Total Score During Double-blind Phase | Baseline, Days 8 ,15 and 25
  BHS is a self-reported measure to assess one's level of negative expectations or pessimism regarding future. It consists of 20 true-false items that examine respondent's attitude over past week by either endorsing a pessimistic statement or denying an optimistic statement; 9 are keyed false and 11 are keyed true. For every statement, each response was assigned score of 0 or 1. Total BHS score is sum of item responses, ranged from 0-20, where higher score represented higher level of hopelessness.
Change From Baseline in Beck Scale for Suicide Ideation -Chinese Version (BSI-CV) Total Score During Double-blind Phase | Baseline, Days 8 ,15 and 25
  BSI-CV is a self-reported measure with 19 items, scored on a 3-point scale (0 to 2). The final score ranges from 0 to 38, with higher scores indicating a greater likelihood of suicide.
Number of Participants With Treatment Emergent Adverse Events (TEAEs)、Vital Signs Abnormalities、Abnormal Electrocardiogram (ECG) Values et al: DB Treatment Phase | up to Day 25
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | up to Day 25
Maximum Plasma Concentration [Cmax] | up to Day 25
plasma elimination half-life [T1/2] | up to Day 25

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - BEIjing AnDing hospital capital medical university, Beijing
  - Beijing AnDing hospital capital medical university, Beijing
  - Beijing Huilongguan Hospital, Beijing
  - The Fourth People's Hospital of Chengdu, Chengdu
  - Hangzhou Seventh People's Hospital, Hangzhou
  - The fourth affiliated hospital of Anhui medical university, Hefei
  - The affiliated Kangning Hospital of Ningbo University, Ningbo
  - Suzhou Guangji Hospital, Suzhou

IPD SHARING:
Plan to Share IPD: No